CLINICAL TRIAL: NCT00242203
Title: Impact of Neoadjuvant Chemotherapy With or Without Zometa on Occult Micrometastases and Bone Density in Women With Locally Advanced Breast Cancer
Brief Title: Evaluation of Chemotherapy Prior to Surgery With or Without Zometa for Women With Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Novartis (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02-0788 / 201104272
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Neoadjuvant; Micrometastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Micrometastasis | interventions — Zoledronic Acid; Epirubicin; Docetaxel; Trastuzumab; Mastectomy, Modified Radical; Mastectomy, Segmental

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zometa (Experimental): Zometa 4 mg IV every 3 weeks for a total of 17 doses. The first treatment will be given at the time of the first chemotherapy treatment and will continue for approximately 1 year.
  Neoadjuvant therapy
  * Epirubicin 75 mg/m2 IV every 21 days for 4 cycles prior to surgery
  * Docetaxel 75 mg/m2 IV every 21 days for 4 cycles prior to surgery
  Surgery - modified radical mastectomy or breast conserving surgery with axillary lymph node dissection
  Adjuvant therapy
  * Epirubicin 75 mg/m2 IV every 21 days for 2 cycles
  * Docetaxel 75 mg/m2 IV every 21 days for 2 cycles
  * All patients who are found to be Her-2 overexpressing by 3+ by ICH for FSH will receive trastuzumab 6 mg/kg IV every 3 weeks for 1 year post surgery
  Radiation therapy - 50-60 Gy in 1.8-2.0 Gy daily fractions to the breast or chest wall. Internal mammary nodes, supraclavicular fossa nodes and axillary nodal basins will receive 45-50 Gy over 5-6 weeks
  Interventions: Drug: Zometa; Drug: Epirubicin; Drug: Docetaxel; Drug: Trastuzumab; Radiation: External beam radiation; Procedure: Modified radical mastectomy or breast conserving surgery with axillary lymph node dissection
- No Zometa (Active Comparator): Neoadjuvant therapy
  * Epirubicin 75 mg/m2 IV every 21 days for 4 cycles prior to surgery
  * Docetaxel 75 mg/m2 IV every 21 days for 4 cycles prior to surgery
  Surgery - modified radical mastectomy or breast conserving surgery with axillary lymph node dissection
  Adjuvant therapy
  * Epirubicin 75 mg/m2 IV every 21 days for 2 cycles
  * Docetaxel 75 mg/m2 IV every 21 days for 2 cycles
  * All patients who are found to be Her-2 overexpressing by 3+ by ICH for FSH will receive trastuzumab 6 mg/kg IV every 3 weeks for 1 year post surgery
  Radiation therapy - 50-60 Gy in 1.8-2.0 Gy daily fractions to the breast or chest wall. Internal mammary nodes, supraclavicular fossa nodes and axillary nodal basins will receive 45-50 Gy over 5-6 weeks
  Interventions: Drug: Epirubicin; Drug: Docetaxel; Drug: Trastuzumab; Radiation: External beam radiation; Procedure: Modified radical mastectomy or breast conserving surgery with axillary lymph node dissection

INTERVENTIONS:
Drug: Zometa
  Other Names: Zoledronic acid
  Arms: Zometa
Drug: Epirubicin
  Other Names: Ellence
Drug: Docetaxel
  Other Names: Taxotere
Drug: Trastuzumab — ONLY for patients that are Her-2 overexpressing by 3+ by ICH for FSH
  Other Names: Herceptin
Radiation: External beam radiation
Procedure: Modified radical mastectomy or breast conserving surgery with axillary lymph node dissection

SUMMARY:
This study is designed to evaluate the impact of Zometa on clearance of bone marrow micrometastases; the protective effect on chemotherapy-induced loss of bone mineral density; and quality of life in women undergoing treatment for locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed primary invasive ductal or invasive lobular breast adenocarcinoma
* Tumor classified as clinically large T2 (2-5 cm), T3, T4 or any T with N1, N2
* Prior malignancies: limited to curatively treated basal or squamous carcinoma of the skin or history of previous malignancies, treated and now > 5 years disease free
* >= 18 years of age
* Normal left ventricular function by echocardiogram or radioventriculogram
* Karnofsky Performance >= 70

Exclusion Criteria:

* No evidence of distant metastasis present by CT, Bone scan, or physical exam
* If the bone scan or CT scans demonstrate indeterminate lesions, the nature of these lesions may be further clarified by additional testing such as PET or MRI
* No current treatment with Zometa or other bisphosphonates
* No serious functional disorders of the liver or kidneys:
* Serum Creatinine <=2
* ALT/AST/ALK Phos <= 1.5 x upper limit of institutional normal.
* Bili <= 1.5 x upper limit of institutional normal.
* Currently not pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2002-10; Primary Completion 2007-08 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the impact of Zometa (zoledronic acid) on the clearance of bone marrow micrometastases | Prior to therapy initiation, after completion of neoadjuvant chemotherapy, and 12-15 months from registration
Evaluate the protective effect of Zometa (zoledronic acid) on chemotherapy-induced loss of bone mineral density | Prior to therapy initiation and 12-15 months from registration

SECONDARY OUTCOMES:
Impact of Zometa (zoledronic acid) on time and site of relapse | 5 years from registration
Effect of treatment on quality of life in women undergoing treatment for LABC. | Baseline and 12-15 months from registration

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Aft, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Consensus development conference: diagnosis, prophylaxis, and treatment of osteoporosis. Am J Med. 1993 Jun;94(6):646-50. doi: 10.1016/0002-9343(93)90218-e. No abstract available. PMID 8506892
- [Background] Cooper C. The crippling consequences of fractures and their impact on quality of life. Am J Med. 1997 Aug 18;103(2A):12S-17S; discussion 17S-19S. doi: 10.1016/s0002-9343(97)90022-x. PMID 9302893
- [Background] Schurch MA, Rizzoli R, Mermillod B, Vasey H, Michel JP, Bonjour JP. A prospective study on socioeconomic aspects of fracture of the proximal femur. J Bone Miner Res. 1996 Dec;11(12):1935-42. doi: 10.1002/jbmr.5650111215. PMID 8970896
- [Background] Pfeilschifter J, Diel IJ. Osteoporosis due to cancer treatment: pathogenesis and management. J Clin Oncol. 2000 Apr;18(7):1570-93. doi: 10.1200/JCO.2000.18.7.1570. PMID 10735906
- [Background] Cann CE, Martin MC, Genant HK, Jaffe RB. Decreased spinal mineral content in amenorrheic women. JAMA. 1984 Feb 3;251(5):626-9. PMID 6690836
- [Background] Shapiro CL, Manola J, Leboff M. Ovarian failure after adjuvant chemotherapy is associated with rapid bone loss in women with early-stage breast cancer. J Clin Oncol. 2001 Jul 15;19(14):3306-11. doi: 10.1200/JCO.2001.19.14.3306. PMID 11454877
- [Background] Young DM, Fioravanti JL, Olson HM, Prieur DJ. Chemical and morphologic alterations of rabbit bone induced by adriamycin. Calcif Tissue Res. 1975 Jul 4;18(1):47-63. doi: 10.1007/BF02546226. PMID 1148891
- [Background] Glackin CA, Murray EJ, Murray SS. Doxorubicin inhibits differentiation and enhances expression of the helix-loop-helix genes Id and mTwi in mouse osteoblastic cells. Biochem Int. 1992 Oct;28(1):67-75. PMID 1280141
- [Background] Reid IR. Glucocorticoid osteoporosis--mechanisms and management. Eur J Endocrinol. 1997 Sep;137(3):209-17. doi: 10.1530/eje.0.1370209. PMID 9330580
- [Background] Van Staa T, Abenhaim L, Cooper C: Use of cyclic etidronate and prevention of fractures. Bone 20:103s (abstract), 1997
- [Background] Black DM, Cummings SR, Karpf DB, Cauley JA, Thompson DE, Nevitt MC, Bauer DC, Genant HK, Haskell WL, Marcus R, Ott SM, Torner JC, Quandt SA, Reiss TF, Ensrud KE. Randomised trial of effect of alendronate on risk of fracture in women with existing vertebral fractures. Fracture Intervention Trial Research Group. Lancet. 1996 Dec 7;348(9041):1535-41. doi: 10.1016/s0140-6736(96)07088-2. PMID 8950879
- [Background] McClung MR, Geusens P, Miller PD, Zippel H, Bensen WG, Roux C, Adami S, Fogelman I, Diamond T, Eastell R, Meunier PJ, Reginster JY; Hip Intervention Program Study Group. Effect of risedronate on the risk of hip fracture in elderly women. Hip Intervention Program Study Group. N Engl J Med. 2001 Feb 1;344(5):333-40. doi: 10.1056/NEJM200102013440503. PMID 11172164
- [Background] Reid IR, Brown JP, Burckhardt P, Horowitz Z, Richardson P, Trechsel U, Widmer A, Devogelaer JP, Kaufman JM, Jaeger P, Body JJ, Brandi ML, Broell J, Di Micco R, Genazzani AR, Felsenberg D, Happ J, Hooper MJ, Ittner J, Leb G, Mallmin H, Murray T, Ortolani S, Rubinacci A, Saaf M, Samsioe G, Verbruggen L, Meunier PJ. Intravenous zoledronic acid in postmenopausal women with low bone mineral density. N Engl J Med. 2002 Feb 28;346(9):653-61. doi: 10.1056/NEJMoa011807. PMID 11870242
- [Background] Saarto T, Blomqvist C, Valimaki M, Makela P, Sarna S, Elomaa I. Chemical castration induced by adjuvant cyclophosphamide, methotrexate, and fluorouracil chemotherapy causes rapid bone loss that is reduced by clodronate: a randomized study in premenopausal breast cancer patients. J Clin Oncol. 1997 Apr;15(4):1341-7. doi: 10.1200/JCO.1997.15.4.1341. PMID 9193325
- [Background] Delmas PD, Balena R, Confravreux E, Hardouin C, Hardy P, Bremond A. Bisphosphonate risedronate prevents bone loss in women with artificial menopause due to chemotherapy of breast cancer: a double-blind, placebo-controlled study. J Clin Oncol. 1997 Mar;15(3):955-62. doi: 10.1200/JCO.1997.15.3.955. PMID 9060533
- [Background] Senaratne SG, Pirianov G, Mansi JL, Arnett TR, Colston KW. Bisphosphonates induce apoptosis in human breast cancer cell lines. Br J Cancer. 2000 Apr;82(8):1459-68. doi: 10.1054/bjoc.1999.1131. PMID 10780527
- [Background] Guise TA, Yin JJ, Taylor SD, Kumagai Y, Dallas M, Boyce BF, Yoneda T, Mundy GR. Evidence for a causal role of parathyroid hormone-related protein in the pathogenesis of human breast cancer-mediated osteolysis. J Clin Invest. 1996 Oct 1;98(7):1544-9. doi: 10.1172/JCI118947. PMID 8833902
- [Background] Thomas RJ, Guise TA, Yin JJ, Elliott J, Horwood NJ, Martin TJ, Gillespie MT. Breast cancer cells interact with osteoblasts to support osteoclast formation. Endocrinology. 1999 Oct;140(10):4451-8. doi: 10.1210/endo.140.10.7037. PMID 10499498
- [Background] Hauschka PV, Mavrakos AE, Iafrati MD, Doleman SE, Klagsbrun M. Growth factors in bone matrix. Isolation of multiple types by affinity chromatography on heparin-Sepharose. J Biol Chem. 1986 Sep 25;261(27):12665-74. PMID 3745206
- [Background] Pfeilschifter J, Mundy GR. Modulation of type beta transforming growth factor activity in bone cultures by osteotropic hormones. Proc Natl Acad Sci U S A. 1987 Apr;84(7):2024-8. doi: 10.1073/pnas.84.7.2024. PMID 3494250
- [Background] Yin J, Chirgwin J, Taylor S: Dominant negative blockade of the transforming growth factor beta type II receptor decreases breast cancer mediated osteolysis. Journal of Bone and Mineral Research 11:180, 1996
- [Background] Mundy GR, Yoneda T. Bisphosphonates as anticancer drugs. N Engl J Med. 1998 Aug 6;339(6):398-400. doi: 10.1056/NEJM199808063390609. No abstract available. PMID 9691109
- [Background] Sasaki A, Boyce BF, Story B, Wright KR, Chapman M, Boyce R, Mundy GR, Yoneda T. Bisphosphonate risedronate reduces metastatic human breast cancer burden in bone in nude mice. Cancer Res. 1995 Aug 15;55(16):3551-7. PMID 7627963
- [Background] Hall DG, Stoica G. Effect of the bisphosphonate risedronate on bone metastases in a rat mammary adenocarcinoma model system. J Bone Miner Res. 1994 Feb;9(2):221-30. doi: 10.1002/jbmr.5650090211. PMID 8140935
- [Background] Yoneda T, Sasaki A, Dunstan C, Williams PJ, Bauss F, De Clerck YA, Mundy GR. Inhibition of osteolytic bone metastasis of breast cancer by combined treatment with the bisphosphonate ibandronate and tissue inhibitor of the matrix metalloproteinase-2. J Clin Invest. 1997 May 15;99(10):2509-17. doi: 10.1172/JCI119435. PMID 9153295
- [Background] Yoneda T, Michigami T, Yi B, Williams PJ, Niewolna M, Hiraga T. Actions of bisphosphonate on bone metastasis in animal models of breast carcinoma. Cancer. 2000 Jun 15;88(12 Suppl):2979-88. doi: 10.1002/1097-0142(20000615)88:12+3.0.co;2-u. PMID 10898341
- [Background] Elomaa I, Blomqvist C, Porkka L, Lamberg-Allardt C, Borgstrom GH. Treatment of skeletal disease in breast cancer: a controlled clodronate trial. Bone. 1987;8 Suppl 1:S53-6. PMID 2961355
- [Background] Kanis JA, Powles T, Paterson AH, McCloskey EV, Ashley S. Clodronate decreases the frequency of skeletal metastases in women with breast cancer. Bone. 1996 Dec;19(6):663-7. doi: 10.1016/s8756-3282(96)00285-2. PMID 8968035
- [Background] Conte PF, Latreille J, Mauriac L, Calabresi F, Santos R, Campos D, Bonneterre J, Francini G, Ford JM. Delay in progression of bone metastases in breast cancer patients treated with intravenous pamidronate: results from a multinational randomized controlled trial. The Aredia Multinational Cooperative Group. J Clin Oncol. 1996 Sep;14(9):2552-9. doi: 10.1200/JCO.1996.14.9.2552. PMID 8823335
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Jallouk AP, Paravastu S, Weilbaecher K, Aft RL. Long-term outcome of (neo)adjuvant zoledronic acid therapy in locally advanced breast cancer. Breast Cancer Res Treat. 2021 May;187(1):135-144. doi: 10.1007/s10549-021-06100-2. Epub 2021 Feb 16. PMID 33591469
- [Derived] Aft R, Naughton M, Trinkaus K, Watson M, Ylagan L, Chavez-MacGregor M, Zhai J, Kuo S, Shannon W, Diemer K, Herrmann V, Dietz J, Ali A, Ellis M, Weiss P, Eberlein T, Ma C, Fracasso PM, Zoberi I, Taylor M, Gillanders W, Pluard T, Mortimer J, Weilbaecher K. Effect of zoledronic acid on disseminated tumour cells in women with locally advanced breast cancer: an open label, randomised, phase 2 trial. Lancet Oncol. 2010 May;11(5):421-8. doi: 10.1016/S1470-2045(10)70054-1. Epub 2010 Mar 31. PMID 20362507
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu